CLINICAL TRIAL: NCT00444548
Title: Measurement Of Urethral Function In Healthy Female Volunteers - Evaluation Of The Sensitivity of Urethral Reflectometry Compared To Urethral Pressure Profilometry, Using [S,S]-Reboxetine.
Brief Title: Evaluation of A Novel Methodology in the Assessment of Urethral Function Using [S,S]-Reboxetine in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A6061028
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
Keywords: Equipment; Supplies
MeSH Terms: interventions — O-methyl reboxetine

INTERVENTIONS:
Drug: [S,S]-Reboxetine

SUMMARY:
[S,S]-Reboxetine will be used to evaluate pharmacodynamic changes in urethral function in healthy volunteers using a novel methodology

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects, aged 18-65 years.
* Subjects must be non-pregnant and non-lactating, and be either post menopausal (greater than 1 year without menses), surgically sterilized, or using another acceptable form of contraception.
* Subjects of child bearing potential must have confirmed negative pregnancy tests at screening and prior to commencing all study periods.

Exclusion Criteria:

* Evidence or history of clinically significant disease (including drug allergies, but excluding untreated, asymptomatic,seasonal allergies at time of dosing).
* Subjects with any clinically significant abnormality following review of laboratory data, urinalysis and physical examination.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-05; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Reflectometry measurements at visit 2, 3, 4 , 5, 6 and 7.

SECONDARY OUTCOMES:
Urethral pressure profile measurements at visit 2, 3, 4, 5, 6 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Hellerup, Denmark

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061028&StudyName=Evaluation%20of%20A%20Novel%20Methodology%20in%20the%20Assessment%20of%20Urethral%20Function%20Using%20%5BS%2CS%5D-Reboxetine%20in%20healthy%20volunteers